CLINICAL TRIAL: NCT01720056
Title: Assessment of Verapamil as an Adjunct for Prevention of Keloid Recurrence After Surgical Removal
Brief Title: Verapamil vs Steroid to Prevent Keloid Recurrence
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Objective of study achieved after interim analysis.
Sponsor: The University of Western Australia (Other)
Responsible Party: Principal Investigator, Fiona M. Wood, Prof. Wood, The University of Western Australia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EC 067/2012
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Keloid Scars
MeSH Terms: conditions — Keloid | interventions — Verapamil; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verapamil (Active Comparator): Verapamil 2.5 mg/mL injection sc intralesionally
  Interventions: Drug: Verapamil
- Kenalog 10 (Active Comparator): Kenalog 10 mg/mL injection sc intralesionally
  Interventions: Drug: Kenalog 10

INTERVENTIONS:
Drug: Verapamil
  Arms: Verapamil
Drug: Kenalog 10
  Arms: Kenalog 10

SUMMARY:
Keloid scarring is a severe cosmetic and painful disease of the skin. The gold standard treatment is yet to be clarified. This randomized clinical pilot study will compare the effects of two local treatments for preventing keloid recurrence after surgical removal; steroid and verapamil.

Study hypothesis: Intralesional therapy with the calcium antagonist verapamil has equal treatment efficacy as steroid injection.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing surgical removal of keloid
* Patient 18 years old or greater
* Length of excisional scar after surgical removal of keloid between 2 and 10 cm

Exclusion Criteria:

* Keloid in face or hands
* Pregnancy or lactation
* Dementia
* Any heart or pulmonary condition
* Systemic treatment with beta-blockers, ACE-inhibitors or calcium antagonists
* Systemic corticosteroidal therapy
* Intralesional steroid treatment within 2 months of surgery to remove keloid
* Flap surgery
* Lesions to face, hands and other cosmetically sensitive areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Keloid recurrence | 1 year

SECONDARY OUTCOMES:
Vancouver Scar Scale Score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fiona M Wood, Professor, Principal Investigator — The University of Western Australia
Locations (1):
- Royal Perth Hospital, Perth, Western Australia, Australia